CLINICAL TRIAL: NCT07335731
Title: Study on the Safety and Efficacy of Domestic Single-Port Robot-Assisted Metabolic Bariatric Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hua Meng, Director of the General Surgery Department & Obesity and Metabolic Disease Center of China-Japan Friendship Hospital, China-Japan Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-HX-177
Record Dates: First submitted 2025-11-15; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Robot Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic surgical treatment group (Experimental)
  Interventions: Device: Robot-assisted single-port bariatric surgery

INTERVENTIONS:
Device: Robot-assisted single-port bariatric surgery — For overweight or obese patients (BMI≥27.5kg/m2) who meet the indications for metabolic surgery, single-port robot-assisted sleeve gastrectomy or gastric bypass surgery is performed.

SUMMARY:
This study aims to obtain short-term clinical results on the safety and efficacy of single-port robot-assisted metabolic weight loss surgery, and to provide further evidence for the clinical promotion of single-port robot systems.

ELIGIBILITY:
Inclusion Criteria:

* ①Overweight or obese patients who meet the criteria for metabolic weight loss surgery, with a BMI ≥ 27.5 kg/m2; ② Patients who understand the purpose of the trial, voluntarily participate in the trial, and sign an informed consent form.

Exclusion Criteria:

* ① Patients who cannot tolerate general anesthesia, such as those with severe heart, lung, or liver dysfunction; ② Patients with severe coagulation disorders; ③ Pregnant patients; ④ Patients with concurrent tumors; ⑤ Patients with extensive and severe abdominal adhesions that prevent the establishment of pneumoperitoneum; ⑥ A BMI > 50 kg/m² is a relative contraindication; ⑦ Patients deemed unsuitable for participation in this trial by any other investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of weight loss | Postoperative 1 month, 3 months, 6 months, 12months

SECONDARY OUTCOMES:
blood pressure | 1 month, 3 months, 6 months, and 12 months post-surgery
operation time | Intraoperative
Postoperative complications (postoperative bleeding, gastric leakage, anastomotic leakage, abdominal infection, incisional hernia, etc.) | 12 months post-surgery
Physician fatigue level (Visual Analogue Scale) | 1 day after surgery
blood sugar | 1 month, 3 months, 6 months, and 12 months post-surgery
body fat percentage | 1 month, 3 months, 6 months, and 12 months post-surgery
estimated blood loss | 1 month after surgery
conversion to laparoscopic or open surgery | 1 month after surgery
30-day reoperation rate | 1 month after surgery
30-day readmission rate | 1 month after surgery
length of postoperative hospital stay | 1 month after surgery
Physician satisfaction level (Net Promoter Score, NPS) | 1 day after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China